CLINICAL TRIAL: NCT04197492
Title: A Phase II Study of Hypofractionated Stereotactic Radiotherapy Combined With Anlotinib in Patients With Recurrent High-Grade Glioma
Brief Title: Hypofractionated Stereotactic Radiotherapy With Anlotinib in Patients With Recurrent High-Grade Gliomas
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Huashan Hospital (Other)
Responsible Party: Principal Investigator, Chongbo Zhao, Head of CyberKnife Center, Principal Investigator, Huashan Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: KY2019-525; HSCK-002 (Other: CyberKinfe Center, Huashan Hospital)
Record Dates: First submitted 2019-12-11; First posted 2019-12-13 (Actual); Last update posted 2024-01-05 (Actual); Status verified 2024-01

CONDITIONS: Malignant Glioma
Keywords: Hypofractionated Stereotactic Radiotherapy; Recurrent High-grade Glioma; Anlotinib
MeSH Terms: conditions — Glioma | interventions — anlotinib

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (1):
- HSRT With Anlotinib (Experimental): * Hypofractionated stereotactic radiotherapy using CyberKnife 25Gy/5fx, 5 days a week for 1 week.
  * Anlotinib once daily (12mg/d) orally administered on days 1-14 of a 21-day cycle until disease progression or treatment intolerance.
  Interventions: Radiation: Hypofractionated Stereotactic Radiotherapy; Drug: Anlotinib

INTERVENTIONS:
Radiation: Hypofractionated Stereotactic Radiotherapy — Hypofractionated stereotactic radiotherapy (CyberKnife, 25Gy/5fx)
  Other Names: Hypofractionated Stereotactic Radiosurgery
Drug: Anlotinib — Anlotinib once daily (12mg/d) on days 1-14 of a 21-day cycle.
  Other Names: AL3818

SUMMARY:
A Phase II Study of Hypofractionated Stereotactic Radiotherapy (HSRT) With Anlotinib in Patients With Recurrent High-Grade Glioma. The primary endpoint is overall survival after radiotherapy. Secondary endpoints included progress-free survival, objective response rate, cognitive function, quality of life, toxicity.

DETAILED DESCRIPTION:
Original histopathologically proven diagnosis World Health Organization (WHO) Grade 3/4 glioma patients who underwent surgery, chemoradiotherapy and adjuvant chemotherapy (Stupp Protocol). Recurrence based on Response Assessment in Neuro-Oncology (RANO) criteria and/or histopathology. Intervention included CyberKnife hypofractionated stereotactic radiotherapy (25Gy/5fx) with Anlotinib once daily (12mg/d) on days 1-14 of a 21-day cycle.

ELIGIBILITY:
Inclusion Criteria:

1. 18-70 years of age;
2. Karnofsky performance status (KPS) ≥ 60;
3. Original histopathologically proven diagnosis World Health Organization (WHO) Grade 4 glioma;
4. Underwent surgery, chemoradiotherapy and adjuvant chemotherapy (Stupp Protocol) after initial diagnosis, recurrent based on the Response Assessment in Neuro-Oncology (RANO) criteria and/or histopathologically proven;
5. Measurable disease;
6. Estimated survival of at least 3 months;
7. Hgb > 9 gm; absolute neutrophil count (ANC) > 1500/μl; platelets > 100,000; Creatinine < 1.5 times the upper limit of laboratory normal value; Bilirubin < 2 times the upper limit of laboratory normal value; serum glutamate pyruvate transaminase (SGPT) or serum glutamate oxaloacetate transaminase (SGOT) < 3 times the upper limit of laboratory normal value;
8. Signed informed consent form;
9. Agreed to participate the follow-up.

Exclusion Criteria:

1. Prior invasive malignancy unless disease free;
2. Received re-irradiation;
3. More than 3 relapses or evidence of subtentorial recurrent disease or tumor greater than 6 cm in maximum diameter;
4. Prior therapy with an inhibitor of vascular endothelial growth factor (VEGF) or VEGFR;
5. Pregnancy or or nursing mothers;
6. Participated in other trials after diagnosis of recurrent;
7. Influence factors toward oral medications;
8. Patients with CTCAE5.0 grade 3+ bleeding;
9. Suffering from severe cardiovascular disease: myocardial ischemia or myocardial infarction above grade II, poorly controlled arrhythmias (including men with QTc interval ≥ 450 ms, women ≥ 470 ms); according to NYHA criteria, grades III to IV Insufficient function, or cardiac color Doppler ultrasound examination indicates left ventricular ejection fraction (LVEF) <50%;
10. Long-term unhealed wounds or fractures;
11. History of organ transplantation;
12. Serious diseases that endanger patients' safety or affect patients' completion of research,according to the researchers' judgment.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 22 (Estimated)
Dates: Start 2019-12-16 (Actual); Primary Completion 2023-12-31 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
Overall survival (OS) | From the start of treatment to the date of death or the last follow-up, up to approximately 24 months
  Estimated using the Kaplan-Meier method

SECONDARY OUTCOMES:
Progression-free survival (PFS) | From the start of treatment to the date of disease progression or death, up to approximately 24 months
  Estimated using the Kaplan-Meier method
Objective response rate (ORR) | Bimonthly up to intolerance the toxicity or progressive disease (PD), up to approximately 24 months
  ORR is defined as the percentage of subjects with evidence of a confirmed complete response (CR) or partial response (PR) as per Response Assessment in Neuro-Oncology (RANO) prior to progression or any further therapy.
Quality of Life score (QoL): European Organization for the Research and Treatment of Cancer Quality of Life Questionnaire (EORTC QLQ-C30) version 3.0 | Bimonthly up to intolerance the toxicity or PD, up to approximately 24 months
  EORTC QLQ-C30 (version 3.0) questionnaire to evaluate the quality of life. All scales range in score from 0 to 100. A high score for a functional scale represents a high / healthy level of functioning, a high score for the global health status / QoL represents a high QoL, but a high score for a symptom scale / item represents a high level of symptomatology / problems.
Cognitive function | Bimonthly up to intolerance the toxicity or PD, up to approximately 24 months
  Mini-Mental State Exam (MMSE, score range 0 to 30) to evaluate the cognitive function. Any score of 24 or more (out of 30) indicates a normal cognition. Below this, scores can indicate severe (≤9 points), moderate (10-18 points) or mild (19-23 points) cognitive impairment.
Toxicity rate | Bimonthly up to intolerance the toxicity or PD, up to approximately 24 months
  Common Terminology Criteria for Adverse Events (CTCAE) 5.0 to assess the toxicity. Estimated using an exact binomial distribution together with 95% confidence interval.

CONTACTS AND LOCATIONS:
Overall Officials: Enmin Wang, MD, Principal Investigator — Huashan Hospital
Locations (1):
- CyberKnife Center, Department of Neurosurgery, Huashan Hospital, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Wuthrick EJ, Curran WJ Jr, Camphausen K, Lin A, Glass J, Evans J, Andrews DW, Axelrod R, Shi W, Werner-Wasik M, Haacke EM, Hillman GG, Dicker AP. A pilot study of hypofractionated stereotactic radiation therapy and sunitinib in previously irradiated patients with recurrent high-grade glioma. Int J Radiat Oncol Biol Phys. 2014 Oct 1;90(2):369-75. doi: 10.1016/j.ijrobp.2014.05.034. Epub 2014 Aug 4. PMID 25104067
- [Background] Clarke J, Neil E, Terziev R, Gutin P, Barani I, Kaley T, Lassman AB, Chan TA, Yamada J, DeAngelis L, Ballangrud A, Young R, Panageas KS, Beal K, Omuro A. Multicenter, Phase 1, Dose Escalation Study of Hypofractionated Stereotactic Radiation Therapy With Bevacizumab for Recurrent Glioblastoma and Anaplastic Astrocytoma. Int J Radiat Oncol Biol Phys. 2017 Nov 15;99(4):797-804. doi: 10.1016/j.ijrobp.2017.06.2466. Epub 2017 Jun 30. PMID 28870792
- [Background] Minniti G, Scaringi C, De Sanctis V, Lanzetta G, Falco T, Di Stefano D, Esposito V, Enrici RM. Hypofractionated stereotactic radiotherapy and continuous low-dose temozolomide in patients with recurrent or progressive malignant gliomas. J Neurooncol. 2013 Jan;111(2):187-94. doi: 10.1007/s11060-012-0999-9. Epub 2012 Nov 6. PMID 23129347
- [Derived] Guan Y, Li J, Gong X, Zhu H, Li C, Mei G, Liu X, Pan L, Dai J, Wang Y, Wang E, Liu Y, Wang X. Safety and Efficacy of Hypofractionated Stereotactic Radiotherapy with Anlotinib Targeted Therapy for Glioblastoma at the First Recurrence: A Preliminary Report. Brain Sci. 2022 Apr 2;12(4):471. doi: 10.3390/brainsci12040471. PMID 35448002